CLINICAL TRIAL: NCT02579213
Title: Examining the Ability of Electronic Nose in Detecting Fetal Chromosomal Disorders
Brief Title: Electronic Nose and Fetal Chromosomal Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0200-15-RMB
Record Dates: First submitted 2015-09-03; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Detecting Abnormal Fetal Karyotype by the Electronic Nose
Keywords: electronic nose; abnormal fetal karyotype
MeSH Terms: interventions — Amniocentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — .33 ml of amniotic fluid are drawn from the uterine cavity, when 30 cc are part of routine tests and the rest of the amount (3 ml) is intended for research

GROUPS / COHORTS (1):
- women candidates for amniocentesis: pregnant women candidates for amniocentesis between 17-33 gestational weeks
  Interventions: Other: observational study done only in women candidate for amniocentesis

INTERVENTIONS:
Other: observational study done only in women candidate for amniocentesis — As a part of routine test in women with obstetrical indication for amniocentesis, we take 30 cc of amniotic fluid. only additional 3 ml of the amniotic fluid are needed for examination by electronic sensors.

SUMMARY:
"electronic nose"- the tiny sensors, will smell and detect the changes in the sample of abnormal fetal karyotype, and fluid that will be confirmed by amniocentesis.

DETAILED DESCRIPTION:
The biochemical engineering department had developed a device called "electronic nose" that can detect various diseases Including cancer and asthma on basis of evaporable substances. The device simulates the human nose ", which includes an array of tiny sensors connected to nanometric sizes electronic calculating unit.. Thanks to their small size, electrical, physical and chemical properties, the sensitive sensors smell and identified changes in composition of the materials that characterize various diseases including kidney disease and asthma.

The electronic nose was developed by Professor Haick from the Technion. The main concept of the device is testing and characterization a trace amounts of substances in the air with the help of nana-technology sensors the idea is revolutionary and would allow the diagnosis of different diseases, like cancer, by exhaling air into the device.

The test is simple and not complicated to perform ,the examiner inhale air into a bag which connected to the "electronic nose". The molecules of the patient's breath will be tied to sensors and transmit an electrical signal to computer chip.

After processing the data the "electronic nose "can distinguish between normal cells and pathological cells.

Hypothesis: the tiny sensors ("electronic nose") will smell and detect the changes in the sample of abnormal fetal karyotype, and fluid that will be confirmed by amniocentesis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women candidates for amniocentesis
* 17-33 gestational weeks

Exclusion Criteria:

* women that refuse to participate in the research
* women older than 45 or less than 16

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A prospective study that includes pregnant women candidates for amniocentesis between 17-33 gestational weeks
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Examining the ability of the electronic nose in detecting abnormal fetal karyotype | 3 years
  the electronic nose can detect various diseases Including cancer and asthma on basis of evaporable substances. The device simulates the human nose ", which includes an array of tiny sensors connected to nanometric sizes electronic calculating unit.
  30 cc of amniotic fluid are part of routine tests and the rest of the amount (3 ml) is intended for research, this sample will be saved in cooling (-20) and subsequently transferred to the Technion, for examination by electronic sensors. The amount of amniotic fluid designed for research is a minimal amount and will not hurt the fetus. At the end of the study following the data processing, we will be able to appreciate the effectiveness of the electronic nose in diagnosing fetal chromosomal disorders.